CLINICAL TRIAL: NCT05225584
Title: A Phase 1, Multicenter, Open-Label, Dose-Escalation and Expansion Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of Intravenously Administered KT-333 in Adult Patients With Relapsed or Refractory Lymphomas, Large Granular Lymphocytic Leukemia, and Solid Tumors
Brief Title: Safety, PK, PD, Clinical Activity of KT-333 in Adult Patients With Refractory Lymphoma, Large Granular Lymphocytic Leukemia, Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kymera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KT333-TL-101
Record Dates: First submitted 2021-12-16; First posted 2022-02-04 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Non Hodgkin Lymphoma (NHL); Peripheral T-cell Lymphoma (PTCL); Cutaneous T-Cell Lymphoma (CTCL); Large Granular Lymphocytic Leukemia (LGL-L); T-cell Prolymphocytic Leukemia (T-PLL); Solid Tumors
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Leukemia, Large Granular Lymphocytic; Leukemia, Prolymphocytic, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Phase 1a Dose Escalation Lymphomas (Experimental): KT-333 dosed IV weekly in 28 day cycles
  Interventions: Drug: KT-333
- Phase 1a Dose Escalation Solid Tumors (Experimental): KT-333 dosed IV weekly in 28 day cycles
  Interventions: Drug: KT-333
- Phase 1b Dose Expansion PTCL (Experimental): KT-333 dosed IV weekly in 28 day cycles
  Interventions: Drug: KT-333
- Phase 1b Dose Expansion CTCL (Experimental): KT-333 dosed IV weekly in 28 day cycles
  Interventions: Drug: KT-333
- Phase 1b Dose Expansion LGL-L (Experimental): KT-333 dosed IV weekly in 28 day cycles
  Interventions: Drug: KT-333
- Phase 1b Dose Expansion Solid Tumor (Experimental): KT-333 dosed IV weekly in 28 day cycles
  Interventions: Drug: KT-333
- Phase 1a Dose Escalation LGL-L (Experimental): KT-333 dosed IV weekly in 28 day cycles
  Interventions: Drug: KT-333
- Phase 1a Dose Escalation T-PLL (Experimental): KT-333 dosed IV weekly in 28 day cycles
  Interventions: Drug: KT-333

INTERVENTIONS:
Drug: KT-333 — KT-333 will be supplied as 10mg/mL concentration frozen solution to be administered intravenously per the protocol defined frequency and dose level.

SUMMARY:
This Phase 1a/1b study will evaluate the safety, tolerability and the pharmacokinetics/pharmacodynamics (PK/PD) of KT-333 in Adult patients with Relapsed or Refractory (R/R) Lymphomas, Large Granular Lymphocytic Leukemia (LGL-L), T-cell prolymphocytic leukemia (T-PLL), and Solid Tumors. The Phase 1a stage of the study will explore escalating doses of single-agent KT-333. The Phase Ib stage will consist of 4 expansion cohorts to further characterize the safety, tolerability and the pharmacokinetics/pharmacodynamics (PK/PD) of KT-333 in Peripheral T-cell Lymphoma (PTCL), Cutaneous T-Cell Lymphoma (CTCL), LGL-L, and solid tumors.

DETAILED DESCRIPTION:
This is an open-label Phase 1a (dose escalation)/1b (dose expansion) first-in-human study of KT-333 in adult patients. Patients with relapsed/refractory (R/R) lymphomas, LGL-L, T-PLL, and solid tumors will be enrolled in Phase 1a. Phase 1b will consist of separate cohorts of patients with R/R PTCL, CTCL, LGL-L, and solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Phase 1a Only: Cytologically or pathologically confirmed Lymphomas (including Hodgkin's, B-cell, T-cell, Small Lymphocytic, or Natural-Killer (NK)-cell Lymphomas and LGL-L), T-PLL and solid tumors with the exception of chronic lymphocytic leukemia (CLL) Note: Patients with indolent non-Hodgkin's lymphoma (NHL) and small lymphocytic lymphoma (SLL) are only eligible if not require immediate cytoreductive therapy or if there are no available treatments with potential benefit.
2. Phase 1b Only: Histologically or pathologically confirmed PTCL, CTCL, LGL-L [T-cell LGL-L or Chronic Lymphoproliferative Disorder of NK-cells (CLPD-NK)], or solid tumors.
3. Fresh or archival formalin fixed paraffin embedded (FFPE) tumor tissue or 15 slides preferably collected within 6 months or 2 years prior to first dose of the study drug (for lymphoma and solid tumor patients respectively).
4. Phase 1a only: Lymphoma and Solid Tumor: Relapsed and/or refractory disease to at least 2 prior systemic standard of care treatments or for whom standard therapies are not available.
5. Phase 1a: LGL-L/T-PLL only: Relapsed and/or refractory disease to at least 1 prior systemic standard of care treatment or for whom standard therapies are not available.
6. Phase 1b only: All disease types: Relapsed and/or refractory disease to at least 1 prior systemic standard of care treatments or for whom standard therapies are not available.
7. LGL-L patients only (hematology specific criteria):

   * One of the following:

     * Severe neutropenia < 500/mm3, or,
     * Symptomatic anemia and/or,
     * Transfusion-dependent anemia.
   * ANC ≥ 200/μL at Screening and C1D1 (pre dose)
   * Platelet count ≥ 100,000/μL (assessed ≥ 7 days following last platelet transfusion in patients with thrombocytopenia requiring platelets).
8. LGL-L Patients Only (baseline disease characteristics):

   * CD3+CD8+ cell population >650/mm3;
   * CD3+CD8+CD57+ population >500/mm3;
   * Presence of a clonal T-cell receptor (within 1 month of diagnosis);
   * Note: patients with T-LGLL may be included with PI approval even if CD3+CD8+ cell population is<650/mm3 or CD3+CD8+CD57+ population is <500/mm3, though +TCR is required;
   * NK LGL is also permitted, provided there is a clonal NK-cell population noted with>500 cells/mm3
9. PTCL and solid tumors Only: Measurable disease at Screening. Solid tumor patients with non-measurable disease are allowed in Phase1a
10. T-PLL: Measurable disease per Lugano and/or atypical T lymphocytes quantifiable by flow cytometry or morphology in the peripheral blood or bone marrow.
11. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at Screening and C1D1 (pre-dose).
12. Adequate bone marrow function at Screening and C1D1 (pre-dose) for all patients except those with LGL-L Adequate liver/kidney organ function at Screening and C1D1 (pre-dose) for all patients.
13. Women of childbearing potential (WOCBP) must agree to use highly effective contraceptive methods for the duration of study treatment and 6 months after the last dose of KT333.

Exclusion Criteria:

1. Known active uncontrolled or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth.

   Note: Patients with solid tumors are eligible if their CNS metastases or cord compression have been treated (e.g., radiotherapy, stereotactic surgery) and they are clinically stable, off steroids for at least 4 weeks before first dose of study drug and have no evidence of progression at time of study enrollment.

   Note: Patients with lymphomas are eligible if their CNS metastases or cord compression have been treated effectively (i.e. achieved CR) and there is no clinical or radiographic evidence of active lymphoma.
2. Diagnosis of Chronic Lymphocytic Leukemia (CLL).
3. History of or active concurrent malignancy other than lymphoma or solid tumors unless the patient has been disease-free for ≥ 2 years.
4. Patient has not recovered from any clinically significant adverse events (AEs) of previous treatments to pretreatment baseline or Grade 1 prior to first dose of study drug.
5. Ongoing unstable cardiovascular function.
6. Autologous hematopoietic stem cell transplant less than 3 months prior to first dose of study drug.
7. Prior allogenic hematopoietic or bone marrow transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Safety | Safety will be assessed from the time ICF signature through 30 days post dose or prior to start of a new anticancer therapy
  Incidence and severity of adverse events as assessed by CTCAE v5.0 Phase 1a/1b
Safety | Safety will be assessed from the time ICF signature through 30 days post dose or prior to start of a new anticancer therapy
  Incidence and severity of clinical laboratory abnormalities in Serum Chemistry, Hematology, Coagulation Parameters and urinalysis tests as assessed by CTCAE v5.0 Phase 1a/1b
Safety | Safety will be assessed from the time ICF signature through 30 days post dose or prior to start of a new anticancer therapy
  Changes in the ECG parameters, including heart rate and measures PR, QRS, QT, and QTc intervals as assessed by CTCAE v5.0 Phase 1a/1b
Maximum Tolerated Dose (MTD) | Within the first 28 days of treatment
  To establish the Maximum Tolerated Dose (MTD) Phase 1a
Dose Limiting Toxicities (DLTs) | Within the first 28days of treatment
  Number of Participants with protocol specified Dose Limiting Toxicities (DLTs) Phase 1a

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve for KT-333 | Blood samples for PK analysis collected at multiple visits during cycle 1 and cycle 2 (each cycle is 28days)
  Area under the plasma concentration versus time curve for KT-333 from time to zero to last quantifiable time point (AUC 0-t ) Phase 1a/1b
Maximum Plasma Concentration of KT-333 (Cmax) | Blood samples for PK analysis collected at multiple visits during cycle 1 and cycle 2 (each cycle is 28days)
  Maximum Plasma Concentration of KT-333 (Cmax)
Time of maximum plasma concentration of KT-333 (Tmax) | Blood samples for PK analysis collected at multiple visits during cycle 1 and cycle 2 (each cycle is 28days)
  Time of maximum plasma concentration of KT-333 (Tmax) Phase 1a/1b
Half-life of KT-333 if data permits (T1/2) | Blood samples for PK analysis collected at multiple visits during cycle 1 and cycle 2 (each cycle is 28days)
  Half-life of KT-333 if data permits (T1/2) Phase 1a/1b
Amount of KT-333 dose excreted in urine from time zero to last collected time point (Ae0-t) | Urine samples for PK analysis collected at multiple visits during cycle 1 and cycle 2 (each cycle is 28days)
  Amount of KT-333 dose excreted in urine from time zero to last collected time point (Ae0-t) Phase 1a
Evidence of clinical activity of KT-333 | From date of baseline scan until the date of first documented progression or date of death from any cause, whichever came first, about 18 months
  Evidence of clinical activity of KT-333 as determined by Objective Response Rate (ORR) as per Lugano criteria 2014 for Lymphomas Phase 1a/1b.
Evidence of clinical activity of KT-333 | From date of baseline scan until the date of first documented progression or date of death from any cause, whichever came first, about 18 months
  Evidence of clinical activity of KT-333 as determined by RECIST 1.1 to determine ORR , complete response (CR), partial response (PR) for solid tumors Phase 1a/1b.
Evidence of clinical activity of KT-333 | Composite assessment from date of baseline assessment until the date of first documented progression or date of death from any cause, whichever came first, about 18 months
  Evidence of clinical activity of KT-333 as determined by ORR by Modified Severity-Weighted Assessment Tool (mSWAT) for Cutaneous T-Cell Lymphoma (CTCL) Phase 1a/1b
Evidence of clinical activity of KT-333 | From date of baseline scan until the date of first documented progression or date of death from any cause, whichever came first, about 18 months
  Evidence of clinical activity of KT-333 as determined by ORR by investigator assessment for Large Granular Lymphocytic Leukemia (LGL-L) Phase 1a/1b
Evidence of clinical activity of KT-333 | From date of baseline scan until the date of first documented progression or date of death from any cause, whichever came first, about 18 months
  Evidence of clinical activity of KT-333 as determined by ORR based on T-PLL International Study Group criteria, Phase 1a
Duration of Response (DOR) | From date of first of response to the date of documented first progression or death whichever comes first, about 18 months
  Duration of Response (DOR) Phase 1a/1b

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Gollerkeri, MD, Study Director — Kymera Therapeutics, Inc.
Locations (13):
- United States (13):
  - UC Irvine Health-Chao Family Comprehensive Cancer Center, Orange, California
  - Norton Cancer Institute, Louisville, Kentucky
  - Henry Ford Hospital, Detroit, Michigan
  - Hackensack University Medical Center, John Theurer Cancer Center, Hackensack, New Jersey
  - Montefiore Medical Center, The University Hospital for Albert Einstein College of Medicine, The Bronx, New York
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Abramson Cancer Center of the University of Pennsylvania Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Emily Couric Cancer Center, Charlottesville, Virginia
  - University of WA/Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No